CLINICAL TRIAL: NCT05631704
Title: A Phase 1 Double-Blind (Sponsor-unblinded), Placebo-Controlled Randomized, Single and Multiple Ascending Dose First-Time-in-Human Study to Investigate the Safety, Tolerability, and Pharmacokinetics of VH4524184 and the Potential for Changes in Cytochrome P450 3A (CYP3A) Activity
Brief Title: A Study to Investigate Safety, Tolerability, and Pharmacokinetics (PK) of VH4524184 and the Potential for Changes in Cytochrome P450 3A (CYP3A) Activity
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: ViiV Healthcare (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Treatment
Other Study IDs: 218803
Record Dates: First submitted 2022-11-18; First posted 2022-11-30 (Actual); Last update posted 2025-12-29 (Actual); Status verified 2025-12

CONDITIONS: HIV Infections
Keywords: First-time-in-human; GSK4524184; Healthy volunteers; Multiple Ascending Dose; Single Ascending Dose; VH4524184
MeSH Terms: conditions — HIV Infections | interventions — Midazolam

STUDY DESIGN:
Intervention Model Description: Participants will receive escalating doses of VH4524184 or placebo in Part 1 and Part 2 of the study. In Part 3, participants will receive VH4524184 under fasted and fed conditions.
Who Masked: Participant, Investigator
Masking Description: This will be a double blind study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (19):
- Part 1: Cohort 1: Participants receiving VH4524184 DL1 (Experimental): Eligible participants will receive VH4524184 Dose Level 1 (DL1) during Cohort 1 of Part 1 of the study.
  Interventions: Drug: VH4524184
- Part 1: Cohort 1: Participants receiving Placebo (Placebo Comparator): Eligible participants will receive Placebo matching VH4524184 DL1 during Cohort 1 of Part 1 of the study.
  Interventions: Drug: Placebo
- Part 1: Cohort 2: Participants receiving VH4524184 DL2 (Experimental): Eligible participants will receive VH4524184 DL2 during Cohort 2 of Part 1 of the study.
  Interventions: Drug: VH4524184
- Part 1: Cohort 2: Participants receiving Placebo (Placebo Comparator): Eligible participants will receive Placebo matching VH4524184 DL2 during Cohort 2 of Part 1 of the study.
  Interventions: Drug: Placebo
- Part 1: Cohort 3: Participants receiving VH4524184 DL3 (Experimental): Eligible participants will receive VH4524184 DL3 during Cohort 3 of Part 1 of the study.
  Interventions: Drug: VH4524184
- Part 1: Cohort 3: Participants receiving Placebo (Placebo Comparator): Eligible participants will receive Placebo matching VH4524184 DL3 during Cohort 3 of Part 1 of the study.
  Interventions: Drug: Placebo
- Part 1: Cohort 4: Participants receiving VH4524184 DL4 (Experimental): Eligible participants will receive VH4524184 DL4 during Cohort 4 of Part 1 of the study.
  Interventions: Drug: VH4524184
- Part 1: Cohort 4: Participants receiving Placebo (Placebo Comparator): Eligible participants will receive Placebo matching VH4524184 DL4 during Cohort 4 of Part 1 of the study.
  Interventions: Drug: Placebo
- Part 1: Cohort 5: Participants receiving VH4524184 DL5 (Experimental): Eligible participants will receive VH4524184 DL5 during Cohort 5 (optional) of Part 1 of the study.
  Interventions: Drug: VH4524184
- Part 1: Cohort 5: Participants receiving Placebo (Placebo Comparator): Eligible participants will receive Placebo matching VH4524184 DL5 during Cohort 5 (optional) of Part 1 of the study.
  Interventions: Drug: Placebo
- Part 1: Cohort 6: Participants receiving VH4524184 DL6 (Experimental): Eligible participants will receive VH4524184 DL6 during Cohort 6 (optional) of Part 1 of the study.
  Interventions: Drug: VH4524184
- Part 1: Cohort 6: Participants receiving Placebo (Placebo Comparator): Eligible participants will receive Placebo matching VH4524184 DL6 during Cohort 6 (optional) of Part 1 of the study.
  Interventions: Drug: Placebo
- Part 2: Cohort 7: Participants receiving VH4524184 RL1 (Experimental): Eligible participants will receive VH4524184 Repeat dose Level 1 (RL1) during Cohort 7 (Part 2) of the study.
  Interventions: Drug: VH4524184
- Part 2: Cohort 7: Participants receiving Placebo (Placebo Comparator): Eligible participants will receive Placebo matching VH4524184 RL1 during Cohort 7 (Part 2) of the study.
  Interventions: Drug: Placebo
- Part 2: Cohort 8: Participants receiving VH4524184 RL2 (Experimental): Eligible participants will receive VH4524184 RL2 during Cohort 8 (Part 2) of the study. If Cohort 8 is the highest Part 2 dose cohort, participants may also receive midazolam probe before and following repeat dose administration of VH4524184
  Interventions: Drug: VH4524184; Drug: Midazolam
- Part 2: Cohort 8: Participants receiving Placebo (Placebo Comparator): Eligible participants will receive Placebo matching VH4524184 RL2 during Cohort 8 (Part 2) of the study. If Cohort 8 is the highest Part 2 dose cohort, participants may also receive midazolam probe before and following repeat dose administration of Placebo matching VH4524184.
  Interventions: Drug: Midazolam; Drug: Placebo
- Part 2: Cohort 9: Participants receiving VH4524184 RL3 (Experimental): Eligible participants will receive VH4524184 RL3 during Cohort 9 (Part 2) (optional) of the study. If Cohort 9 is the highest Part 2 dose cohort, participants may also receive midazolam probe before and following repeat dose administration of VH4524184.
  Interventions: Drug: VH4524184; Drug: Midazolam
- Part 2: Cohort 9: Participants receiving Placebo (Placebo Comparator): Eligible participants will receive Placebo matching VH4524184 RL3 during Cohort 9 (Part 2) (optional) of the study. If Cohort 9 is the highest Part 2 dose cohort, participants may also receive midazolam probe before and following repeat dose administration of Placebo matching VH4524184.
  Interventions: Drug: Midazolam; Drug: Placebo
- Part 3: Cohort 10: VH4524184 Fasted/ VH4524184 Fed (Experimental): Eligible participants will receive VH4524184 under fasted condition in Treatment Period 1 followed by VH4524184 under fed condition in Treatment Period 2 during Cohort 10 (Part 3) of the study. Treatment Periods will be separated by a washout period.
  Interventions: Drug: VH4524184

INTERVENTIONS:
Drug: VH4524184 — VH4524184 will be administered.
  Arms: Part 1: Cohort 1: Participants receiving VH4524184 DL1; Part 1: Cohort 2: Participants receiving VH4524184 DL2; Part 1: Cohort 3: Participants receiving VH4524184 DL3; Part 1: Cohort 4: Participants receiving VH4524184 DL4; Part 1: Cohort 5: Participants receiving VH4524184 DL5; Part 1: Cohort 6: Participants receiving VH4524184 DL6; Part 2: Cohort 7: Participants receiving VH4524184 RL1; Part 2: Cohort 8: Participants receiving VH4524184 RL2; Part 2: Cohort 9: Participants receiving VH4524184 RL3; Part 3: Cohort 10: VH4524184 Fasted/ VH4524184 Fed
Drug: Midazolam — Midazolam will be administered in the highest dose cohort in Part 2 (Cohorts 8 or 9).
  Arms: Part 2: Cohort 8: Participants receiving Placebo; Part 2: Cohort 8: Participants receiving VH4524184 RL2; Part 2: Cohort 9: Participants receiving Placebo; Part 2: Cohort 9: Participants receiving VH4524184 RL3
Drug: Placebo — Placebo will be administered.
  Arms: Part 1: Cohort 1: Participants receiving Placebo; Part 1: Cohort 2: Participants receiving Placebo; Part 1: Cohort 3: Participants receiving Placebo; Part 1: Cohort 4: Participants receiving Placebo; Part 1: Cohort 5: Participants receiving Placebo; Part 1: Cohort 6: Participants receiving Placebo; Part 2: Cohort 7: Participants receiving Placebo; Part 2: Cohort 8: Participants receiving Placebo; Part 2: Cohort 9: Participants receiving Placebo

SUMMARY:
This study is designed to investigate the safety, tolerability and PK of VH4524184 (GSK4524184) and the potential of VH4524184 to inhibit or induce CYP3A activity in healthy participants.

ELIGIBILITY:
Inclusion Criteria:

* Participant must be 18 to 50 years of age.
* Participants who are overtly healthy.
* Body weight >=50.0 kilograms (kg) (110 pounds [lbs]) for men and >=45.0 kg (99 lbs) for women and body mass index within the range 18.5 to 32.0 kilograms per meter square (kg/m^2) (inclusive).
* Male or female. Male Participants: No contraceptive restrictions for male participants. Female Participants: A female participant (female sex assigned at birth) is eligible to participate if she is not pregnant, or breastfeeding and is not physically able to have a baby.

Exclusion Criteria:

* History or presence of clinical condition that could significantly alter how medicines are absorbed, broken down or eliminated from the body; be risky to the participant, or make it difficult to interpret the data from the study.
* Pre-existing clinically relevant gastro-intestinal disorders.
* Abnormal blood pressure.
* Certain blood or other cancers within the past 5 years.
* Breast cancer within the past 10 years
* Current or chronic history of liver disease or liver or bile tract abnormalities (with the exception of Gilbert's syndrome or asymptomatic gallstones).
* QT interval corrected for heart rate according to Fridericia's formula (QTcF) >450 milliseconds (msec).
* Medical history of cardiac arrhythmias or cardiac disease or a family and personal history of long QT syndrome.
* History of seizure
* Any known or suspected pre-existing psychiatric condition, including depression, anxiety and insomnia/sleep disturbances.
* Any positive (abnormal) response to the Columbia Suicide Severity Rating Scale (CSSRS).
* Past or intended use of over-the-counter or prescription medication within 7 days (or 14 days if the drug is a potential enzyme inducer) or 5 half-lives (whichever is longer) prior to dosing and for the duration of the study.
* Receipt of any live vaccine(s) or vaccines against Coronavirus disease 2019 (Covid-19) within 28 days prior to screening or plans to receive such vaccines during the study.
* Exposure to more than 4 new investigational products (including long-acting investigational products) within 12 months prior to the first dosing day.
* Current enrollment or past participation in another investigational study in which an investigational intervention (e.g., drug, human blood product, monoclonal antibody, vaccine, invasive device) was administered within the last 30 days, 5 half-lives or twice the duration of the biological effect of the investigational product (whichever is longer) before signing of consent (OR screening) any other clinical study.
* Participation in the study would result in loss of blood or blood products in excess of 500 milliliters (mL) over a 56-day period.
* Current enrollment or past participation in this clinical study.
* Estimated Glomerular Filtration Rate (eGFR) <90 milliliters per minute (mL/min) (calculated using Chronic Kidney Disease Epidemiology Collaboration equation) or serum creatinine >1.1 times Upper limit of normal (ULN).
* Hemoglobin <12.5 grams per deciliter (g/dL) for men and <11 g/dL for women
* ALT or AST >1.5 times ULN
* Total bilirubin >1.5 times ULN (isolated bilirubin >1.5 times ULN is acceptable if bilirubin is fractionated and direct bilirubin <35 percent [%]).
* Any significant arrhythmia or Electrocardiogram (ECG) finding
* Exclusion criteria for Screening ECG (a single repeat is allowed for eligibility determination): Heart rate:<45 or >100 beats per minute (bpm) (Males), <50 or >100 bpm (Females); PR interval: <120 or >220 msec; QRS duration: <70 or >120 msec and QTcF interval: >450 msec.
* Presence of hepatitis B surface antigen (HBsAg) at screening.
* Positive Hepatitis C antibody test result at screening
* Positive pre-study drug/alcohol screen.
* Positive human immunodeficiency virus (HIV) antibody test.
* Regular alcohol consumption within 6 months prior to the study
* Regular use of known drugs of abuse
* Urinary cotinine levels indicative of smoking or history or regular use of tobacco- or nicotine-containing products within 6 months prior to screening and at admission.
* Sensitivity to the study drug, or components thereof, midazolam (For Part 2, midazolam probe cohort), excipients contained therein, benzodiazepines, or other drug or other allergy that, in the opinion of the investigator or Sponsor Medical Monitor, contraindicates participation in the study.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 84 (Actual)
Dates: Start 2022-12-02 (Actual); Primary Completion 2023-07-27 (Actual); Study Completion 2023-07-27 (Actual)

PRIMARY OUTCOMES:
Part 1: Number of participants with serious adverse events (SAE) and non-serious adverse events (non-SAE) | Up to 4 weeks
Part 2: Number of participants with SAE and non-SAE | Up to 6.5 weeks
Part 3: Number of participants with SAE and non-SAE | Up to 6.5 weeks
Part 1: Number of participants with adverse events based on severity | Up to 4 weeks
Part 2: Number of participants with adverse events by severity | Up to 6.5 weeks
Part 3: Number of participants with adverse events based on severity | Up to 6.5 weeks
Part 1: Percentage of participants who discontinue treatment due to adverse events (AE) | Up to 4 weeks
Part 2: Percentage of participants who discontinue treatment due to AE | Up to 6.5 weeks
Part 3: Percentage of participants who discontinue treatment due to AE | Up to 6.5 weeks
Part 1: Change from Baseline in Aspartate aminotransferase (AST), Alanine aminotransferase (ALT) and Alkaline phosphatase (ALP) (International units per liter) | Baseline (Day 1) and up to 4 weeks
Part 2: Change from Baseline in AST, ALT and ALP (International units per liter) | Baseline (Day 1) and up to 6.5 weeks
Part 3: Change from Baseline in AST, ALT and ALP (International units per liter) | Baseline (Day 1) and up to 6.5 weeks
Part 1: Change from Baseline in Total bilirubin and Direct bilirubin (Micromoles per liter) | Baseline (Day 1) and up to 4 weeks
Part 2: Change from Baseline in Total bilirubin and Direct bilirubin (Micromoles per liter) | Baseline (Day 1) and up to 6.5 weeks
Part 3: Change from Baseline in Total bilirubin and Direct bilirubin (Micromoles per liter) | Baseline (Day 1) and up to 6.5 weeks
Part 1: Change from Baseline in Prothrombin time and Partial Thromboplastin Time (Seconds) | Baseline (Day 1) and up to 4 weeks
Part 2: Change from Baseline in Prothrombin time and Partial Thromboplastin Time (Seconds) | Baseline (Day 1) and up to 6.5 weeks
Part 3: Change from Baseline in Prothrombin time and Partial Thromboplastin Time (Seconds) | Baseline (Day 1) and up to 6.5 weeks
Part 1: Change from Baseline in International normalized ratio (INR) (Ratio) | Baseline (Day 1) and up to 4 weeks
Part 2: Change from Baseline in INR (Ratio) | Baseline (Day 1) and up to 6.5 weeks
Part 3: Change from Baseline in INR (Ratio) | Baseline (Day 1) and up to 6.5 weeks
Part 1: Number of participants with maximum toxicity grade increase from Baseline in liver panel laboratory parameters; AST, ALT, ALP, Total bilirubin, Direct bilirubin, Prothrombin time, Partial Thromboplastin Time and INR | Baseline (Day 1) and up to 4 weeks
Part 2: Number of participants with maximum toxicity grade increase from Baseline in liver panel laboratory parameters; AST, ALT, ALP, Total bilirubin, Direct bilirubin, Prothrombin time, Partial Thromboplastin Time and INR | Baseline (Day 1) and up to 6.5 weeks
Part 3: Number of participant with maximum toxicity grade increase from Baseline in liver panel laboratory parameters; AST, ALT, ALP, Total bilirubin, Direct bilirubin, Prothrombin time, Partial Thromboplastin Time and INR | Baseline (Day 1) and up to 6.5 weeks
Part 1: Area under the plasma-concentration time curve from zero (pre-dose) extrapolated to infinite time (AUC[0-infinity]) following dosing of VH4524184 | Up to 4 weeks
Part 2: Area under the plasma concentration-time curve from zero (pre-dose) to the end of the dosing interval at steady state (AUC[0-tau]) following dosing of VH4524184 | Up to 6.5 weeks
Part 1: Maximum observed plasma drug concentration (Cmax) following dosing of VH4524184 | Up to 4 weeks
Part 2: Cmax following dosing of VH4524184 | Up to 6.5 weeks
Part 1: Time to maximum observed plasma drug concentration (tmax) following dosing of VH4524184 | Up to 4 weeks
Part 2: Tmax following dosing of VH4524184 | Up to 6.5 weeks
Part 1: Apparent terminal half-life (t1/2) following dosing of VH4524184 | Up to 4 weeks
Part 2: T1/2 following dosing of VH4524184 | Up to 6.5 weeks

SECONDARY OUTCOMES:
Part 1: Number of participants with treatment emergent Grade 3 or Grade 4 laboratory abnormalities | Up to 4 weeks
Part 2: Number of participants with treatment emergent Grade 3 or Grade 4 laboratory abnormalities | Up to 6.5 weeks
Part 3: Number of participants with treatment emergent Grade 3 or Grade 4 laboratory abnormalities | Up to 6.5 weeks

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — ViiV Healthcare
Locations (1):
- GSK Investigational Site, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to anonymized individual patient-level data (IPD) and related study documents of the eligible studies via the Data Sharing Portal. Details on GSK's data sharing criteria can be found at: https://www.gsk.com/en-gb/innovation/trials/data-transparency/
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Anonymized IPD will be made available within 6 months of publication of primary, key secondary and safety results for studies in product with approved indication(s) or terminated asset(s) across all indications.
Access Criteria: Anonymized IPD is shared with researchers whose proposals are approved by an Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension may be granted, when justified, for up to 6 months.
URL: https://www.gsk.com/en-gb/innovation/trials/data-transparency/

REFERENCES:
- [Derived] Rogg L, Underwood M, Hanan N, Castillo-Mancilla JR, Kahl L, Halliday F, Ghita GL, Jeffrey JL, Byrne S, Onodera T, Horton J, Gartland M. Phase 1 Evaluation of VH4524184, a Third-Generation Integrase Strand Transfer Inhibitor With an Enhanced Resistance Profile. Clin Infect Dis. 2025 Oct 6;81(3):510-520. doi: 10.1093/cid/ciaf135. PMID 40117383